CLINICAL TRIAL: NCT06975280
Title: Implementation, Cultural Adaptation, and Efficacy Evaluation of Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) for Unaccompanied Refugee Minors in Greece
Brief Title: Trauma-Focused Cognitive Behavioral Therapy in Unaccompanied Refugee Minors With PTSD in Greece: An RCT
Acronym: TF-CBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Theodora Anastasiou (Other)
Collaborators: Greek Ministry of Migration and Asylum (Unknown); SOS Children's Villages (Other)
Responsible Party: Sponsor-Investigator, Theodora Anastasiou, PhD Candidate in Clinical Psychology, Panteion University, Panteion University
Organization: Panteion University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 40/4-10-2023
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Post-Traumatic Stress Disorder (PTSD); Depressive Symptoms; Anxiety Symptoms; Somatic Symptoms; Emotional and Behavioral Difficulties
Keywords: Unaccompanied minors; Refugee adolescents; Trauma-Focused Cognitive Behavioral Therapy; TF-CBT; PTSD; Depression; Anxiety; Child trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Medically Unexplained Symptoms | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the TF-CBT intervention group or the Treatment-as-Usual (TAU) control group, and both groups will be assessed at baseline, post-intervention, and 3-month follow-up.
Who Masked: Participant
Masking Description: Participants are blinded to group assignment (intervention vs. control), but investigators, care providers, and outcomes assessors are aware.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (TF-CBT) (Experimental): Participants in this arm will receive a structured therapeutic protocol based on trauma-focused cognitive behavioral therapy (TF-CBT), delivered over 12 weekly or bi-weekly sessions by trained psychologists in accommodation centers and Supported Independent Living (SIL) programs across Greece. The intervention includes psychoeducation, relaxation techniques, affective modulation, cognitive restructuring, development of a trauma narrative and trauma processing, in vivo exposure, and strategies to enhance safety and future planning. The program is specifically adapted for unaccompanied asylum-seeking minors (UAMs) presenting with symptoms of PTSD.
  Interventions: Behavioral: Trauma - Focused Cognitive Behavioral Therapy
- Control group (TAU) (Active Comparator): Participants in this arm will receive the standard support services (Treatment as Usual) provided in the accommodation centers and Supported Independent Living (SIL) programs, including routine clinical management and general psychological support, without engagement in a structured therapeutic framework or participation in the trauma-focused intervention. Access to the regular psychosocial services available to all residents will remain unchanged.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Trauma - Focused Cognitive Behavioral Therapy — TF-CBT is a comprehensive, evidence-based, short-term therapeutic protocol aimed at reducing trauma-related symptoms in children and adolescents aged 3-18. The protocol consists of 12 double sessions conducted with both the child and their caregiver. Developed for children who have experienced sexual abuse and multiple traumas, TF-CBT has since been successfully applied to a variety of traumatic experiences. Core components of the protocol include psychoeducation, relaxation techniques, emotional regulation, cognitive processing, trauma narrative, in vivo exposure, conjoint child/caregiver sessions, and safety planning. The intervention is culturally informed and flexible to meet individual needs. Adjustments have been made in the context of unaccompanied minors (UAMs), where caregiver involvement is not feasible, due to specific circumstances in accommodation centers and Supportin Greece.
  Other Names: Trauma-Focused CBT; TF-CBT
  Arms: Intervention Group (TF-CBT)
Behavioral: Treatment as Usual (TAU) — The Treatment as Usual (TAU) approach involves routine clinical management and psychological support, without the use of a structured therapeutic framework. This intervention consists of general, non-specific support provided by clinical staff, including informal counseling and monitoring of the child's psychological well-being. Unlike more structured therapeutic protocols, TAU does not follow a predefined set of interventions or techniques, allowing for a flexible and individualized approach, though lacking the formal therapeutic focus of interventions like TF-CBT.
  Other Names: TAU
  Arms: Control group (TAU)

SUMMARY:
This single-blinded, multicentered, randomized controlled trial aims to evaluate the effectiveness of Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) compared to Treatment-as-Usual (TAU) in reducing post-traumatic stress symptoms among unaccompanied refugee minors (UAMs) residing in accommodation centers and Supported Independent Living (SIL) programs in Greece. Participants aged 15-18 will be randomly assigned to either a TF-CBT intervention group or a TAU control group. The intervention will be delivered by trained psychologists under supervision and culturally adapted to the Greek refugee context. Assessments will occur at baseline, post-intervention, and three months later, using standardized psychometric tools. Secondary outcomes include changes in comorbid psychiatric symptoms (depression, anxiety, somatic symptoms), emotional and behavioral difficulties, and quality of life. The study also investigates potential moderators of treatment response such as age, gender, trauma history, and psychiatric comorbidity.

DETAILED DESCRIPTION:
UAMs are a particularly vulnerable population, facing significant risks due to the compounded effects of trauma, displacement, and lack of family support. The study aims to fill a critical gap in the literature by providing an empirical evaluation of TF-CBT for this population, as no previous studies have utilized an RCT design to assess TF-CBT for UAMs in the Greek context.

Study Objectives and Rationale The primary aim of this study is to empirically validate the effectiveness of TF-CBT for UAMs with PTSD symptoms. Secondary objectives include the adaptation of TF-CBT to the Greek cultural context, the development of guidelines for its implementation, and the provision of professional training for psychologists working with UAMs. The study will also assess the impact of TF-CBT on emotional well-being, PTSD symptoms, and overall mental health. Given the growing refugee population in Greece and the high levels of trauma experienced by UAMs, the need for culturally appropriate and evidence-based mental health interventions is urgent.

Study Design and Methodology The study adopts a single-blinded, randomized controlled trial pre-post design, to compare the intervention group (TF-CBT) with the control group (TAU) and assess the efficacy of TF-CBT in accommodation centers and Supported Independent Living (SIL) programs in Greece for UAMs. Effectiveness will be evaluated through within-group comparisons of pre-treatment and post-treatment outcomes for the intervention group, as well as between-group comparisons of the TF-CBT group (n = 30) and the TAU group (n = 30). It is a multicenter study conducted across multiple refugee accommodation centers and Supported Independent Living (SIL) programs throughout Greece. Participants will be randomly assigned to either the intervention group (TF-CBT) or the control group (TAU). The trial will be conducted at three key time points: baseline (T0), immediately after the intervention (T1), and three months post-intervention (T2). Data will be collected through structured questionnaires, including the Child and Adolescent Trauma Screen (CATS) to evaluate trauma exposure and PTSD symptomatology, the Depression, Anxiety, and Stress Scale - 21 items (DASS-21) to measure levels of depressive, anxious, and stress-related symptoms, the Patient Health Questionnaire - 15 (PHQ-15) to assess somatic symptoms, the Strengths and Difficulties Questionnaire (SDQ) to evaluate emotional and behavioral difficulties and the World Health Organization - Five Well-Being Index (WHO-5) to assess overall emotional well-being and quality of life. All tools will be administered in languages familiar to the participants. Official or validated translations will be used when available. These include Greek, English, French, Arabic, Urdu, and Somali. Where validated translations are unavailable, community-based translation and back-translation procedures (Beaton et al., 2000) will be applied, with the assistance of trained volunteer interpreters to ensure cultural and linguistic appropriateness.

While psychologists will oversee the assessment process to ensure it remains supportive and non-intrusive, they will not have access to the assessment data or results. Interpreters will be present when required to facilitate understanding, but they will not participate in the assessment itself. All responses will be anonymized and used solely for the purpose of evaluating the intervention's effectiveness.

Psychologists, who are employed by the accommodation centers and Supported Independent Living (SIL) programs, will also be randomly assigned to the intervention or the control group. Therapists of the intervention group will receive specialized training in TF-CBT prior to the start of the study to ensure the highest quality of treatment and they will administer TF-CBT intervention under supervision. The TAU approach involves minimal intervention, consisting of routine clinical management and psychological support without a structured therapeutic framework. Moreover, the study will be conducted in collaboration with trained interpreters, to ensure that language barriers do not hinder the delivery and evaluation of the intervention.

Demographic Data and Inclusion Criteria Participants in the study will be UAMs aged 15-18 years, currently residing in accommodation centers and Supported Independent Living (SIL) programs in Greece. To be eligible for inclusion, participants should have arrived in Greece as unaccompanied minors, be within the specified age range (15-18 years), have a formal diagnosis of Post-Traumatic Stress Disorder (PTSD) according to DSM-5 criteria, or present with moderate to high levels of traumatic distress as indicated by the Child and Adolescent Trauma Screen (CATS), have maintained a stable living arrangement for at least 2-3 weeks prior to the intervention, and not be scheduled for relocation or transfer within the upcoming 2-3 months following the intervention's initiation. Exclusion criteria include: Diagnosed intellectual disability (IQ < 70) or other developmental disorders that may hinder participation, acute suicidality or recent severe self-injurious behavior, significant risk of violence toward others, comorbidity with bipolar disorder or psychotic disorders, and ongoing substance abuse or active addiction.

Demographic information collected at baseline from both participants and the psychologists delivering the intervention will include age, gender, country of origin, and native language.

Power Analysis The sample size for this study was determined based on an a priori power analysis conducted using G*Power software. A two-tailed t-test for independent samples, with equal group sizes, was selected as the statistical test. The significance level (α) was set at 0.05, and the desired statistical power was 0.80, consistent with standard practice.

The analysis indicated that, for an effect size (d) of 0.75, a minimum of 29 participants per group would be required to achieve satisfactory power. Given this calculation, a sample size of 30 children per group was determined to provide adequate statistical power (1-β) to detect meaningful differences between groups at the specified effect size.

Data Collection and Statistical Analysis Data collection will be conducted electronically using Google Forms, ensuring full confidentiality and participant anonymity. All responses will be anonymized and utilized to evaluate the effectiveness of the intervention across assessment time points.

Statistical analysis will be conducted using SPSS latest edition. Descriptive statistics will summarize the key variables, and independent t-tests and chi-square tests will assess baseline equivalence between the groups. To evaluate the effectiveness of the intervention, a repeated measures ANOVA will examine the interaction between group (intervention vs. control) and time (pre-intervention, post-intervention, and follow-up). Effect size calculations (partial eta-squared and Cohen's d) will be used to quantify the magnitude of observed effects.

Ethical Considerations The study will be conducted in full compliance with the Declaration of Helsinki and has received ethical approval from the Ethics Review Board of Panteion University in Athens, Greece. All participant data will be handled in accordance with the General Data Protection Regulation (GDPR). Prior to participation, all participants will provide informed consent, and psychologists will ensure that the process is voluntary and anonymous. To protect participants' confidentiality, a personal identification code will be used to link responses across time points without collecting personal identifiable information. Data will be securely stored and only accessible by the researchers involved in the study.

Challenges and Limitations Conducting RCTs in refugee populations presents unique challenges, such as limited resources, high mobility of participants, and logistical constraints. The transient nature of UAMs necessitates short follow-up periods, which may limit the ability to assess long-term outcomes. Additionally, cultural and language barriers may affect the implementation and interpretation of both the intervention and assessment tools. However, this study will address these issues using culturally adapted tools, translator verification, and flexible intervention protocols.

Expected Outcomes and Impact The study is expected to provide valuable insights into the effectiveness of TF-CBT for UAMs, contributing to the development of evidence-based guidelines and best practices for treating PTSD in this population. By improving mental health outcomes and offering training for psychologists, the study aims to enhance the quality of care for UAMs in Greece and other refugee-hosting countries. Furthermore, the findings will inform future research on trauma-focused interventions for refugee populations, with the potential for broader application across Europe and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Be unaccompanied upon arrival in Greece and aged between 15-18 years old.
* Being diagnosed with PTSD based on DSM-5 criteria. Young refugees with post-traumatic stress symptoms (PTSS), as delineated by high or moderate trauma-related distress in the Child and Adolescent Trauma Screen (CATS), will also be eligible to participate in the study.
* Reside in an accommodation center or SIL program for UAMs in Greece.
* Have a stable living arrangement for at least 2-3 weeks prior to the intervention.
* Not be expected to relocate within the 2-3 months following the start of the intervention.

Exclusion Criteria:

* a diagnosed intellectual disability (IQ < 70) or another developmental disorder
* acute suicidality or life-threatening self-harm behavior
* significant risk of harm to others
* comorbidity with bipolar disorder or a psychotic disorder
* substance abuse.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Child and Adolescent Trauma Screen (CATS) | Initial assessment (baseline), assessment immediately following the intervention, and a follow-up assessment 3 months after the intervention.
  A standardized measure used to assess trauma-related symptoms in children and adolescents. This tool is used as the primary outcome to evaluate changes in trauma symptoms following the intervention.

SECONDARY OUTCOMES:
DASS-21: Depression, Anxiety, and Stress Scale | Initial assessment (baseline), assessment immediately following the intervention, and a follow-up assessment 3 months after the intervention.
  A 21-item scale used to assess levels of depression, anxiety, and stress. It serves as a secondary outcome to measure emotional distress in participants.
Strengths and Difficulties Questionnaire (SDQ) | Initial assessment (baseline), assessment immediately following the intervention, and a follow-up assessment 3 months after the intervention.
  A behavioral screening tool for children and adolescents that measures emotional symptoms, conduct problems, hyperactivity, peer relationship problems, and prosocial behavior. This will be used to assess general mental health and behavior.
PHQ-15: Physical Health Questionnaire | Initial assessment (baseline), assessment immediately following the intervention, and a follow-up assessment 3 months after the intervention.
  A questionnaire that measures physical symptoms related to health conditions. It will help evaluate any physical health-related outcomes from the intervention.
WHO-5 Well-Being Index | Initial assessment (baseline), assessment immediately following the intervention, and a follow-up assessment 3 months after the intervention.
  A 5-item index used to measure subjective well-being. This tool will assess overall psychological well-being and life satisfaction as a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Vasiliki Yotsidi, PhD, Study Chair — Panteion University
Locations (1):
- General Secretariat for Vulnerable Persons and Institutional Protection, Ministry of Migration and Asylum, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided